CLINICAL TRIAL: NCT04706559
Title: Efficacy of Oral Supplementation of Probiotics in Children With Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Collaborators: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Kamala Acharya, Junior Resident, Department of Dermatology and Venereology, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRC/1886/020; 720/2020 MT (Other: Nepal Health Research Council)
Record Dates: First submitted 2021-01-04; First posted 2021-01-13 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2020-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Lacteol

STUDY DESIGN:
Intervention Model Description: Assessor blinded, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: In this study, there will be three investigators i.e, one principal investigator, and two co-investigators. Among them, one of the co-investigators will be blinded who will act as an assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Interventional group) (Experimental): Along with below mentioned conventional treatment, the participants in group A (i.e. Interventional group) will receive conventional treatment of AD for a short duration along with probiotics for 8 weeks. One probiotic sachet twice a day will be prescribed. A sachet of 2 grams containing 1.25 billion cells per gram of 4 strains (Lactobacillus rhamnosus, Lactobacillus acidophilus, Bifidobacterium longum, and Saccharomyces boulardii) will be used. The child will receive a total of 5 billion cells of probiotics per day.
  Interventions: Drug: Probiotic sachet containing mixture of four strains i.e.Lactobacillus rhamnosus, Lactobacillus acidophilus, Bifidobacterium longum, and Saccharomyces boulardii; Drug: Conventional treatment
- Group B (Conventional group) (Active Comparator): All patients (i.e. in both arms) with atopic dermatitis will be prescribed emollients and cleanser as a part of routine skin care. Topical corticosteroid (i.e. Fluticasone 0.05% cream) and topical calcineurin inhibitor (tacrolimus 0.1% ointment) for sensitive areas like periorbital regions, flexures and face, will be given once daily. All patients will be given an oral antihistamine (syrup/ tablet cetirizine 0.3mg/kg) at night. It is referred to as conventional treatment.
  Interventions: Drug: Conventional treatment

INTERVENTIONS:
Drug: Probiotic sachet containing mixture of four strains i.e.Lactobacillus rhamnosus, Lactobacillus acidophilus, Bifidobacterium longum, and Saccharomyces boulardii — Interventional group: Children with AD meeting eligibility criteria receiving probiotics and conventional treatment (topical corticosteroid, topical tacrolimus, an oral antihistamine and emollients).
  Arms: Group A (Interventional group)
Drug: Conventional treatment — topical corticosteroid, topical tacrolimus, an oral antihistamine and emollients as per atopic dermatitis treatment guidelines.

SUMMARY:
Various clinical studies have evaluated the role of probiotics in children with atopic dermatitis, with some studies showing improvement in clinical outcome after supplementation of probiotics and others showing no additional benefit. This study is to provide clinical evidence of effect of a mixture of probiotics in Atopic Dermatitis (AD) patients based on improvement in SCORAD (SCORing Atopic Dermatitis) index.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is the common chronic inflammatory skin disease with relapsing courses that often start in infancy and childhood. It is characterized by erythema, itchy papules, occasionally vesicles (in infants), which may become excoriated and lichenified and have a typical flexural distribution. Atopy is defined as a "personal or familial tendency to produce immunoglobulin antibodies in response to even low doses of allergen, and associated with development of AD, asthma and rhinoconjunctivitis.The worldwide prevalence of AD is estimated to be 20% in children and 2-10% in adults. The incidence of AD has increased by 2 to 3 folds in past 3 decades in the industrialized countries and represents a major public health burden. According to the International Study of Asthma and Allergies in Childhood (ISAAC) phase 3, the prevalence of AD among the age group of 13 to 14 in Africa and Latin America was at 12-14% and 6-10% respectively. The Asian Pacific countries, the Eastern Mediterranean region and the Indian subcontinent, it was 3-6% among the same age groups (13-14 years). Whereas among 6 to 7 years children, for Asian Pacific countries, Africa and Latin America the prevalence of AD was around 10% and in Indian subcontinent and Eastern Mediterranean region, value was lower at 3-5%

In Nepal the frequency of AD in all age group was 2% as per a year hospital based study done by Singh S and Agrawal S et.al in 2012. (Unpublished data, on personal communication)

The pathogenesis of AD appears to result from interaction between various genetic and environmental factors. It is associated with skin barrier dysfunction and immune dysregulation. The barrier dysfunction is early feature of AD which may be a primary but may also be a secondary to skin inflammation. Lack of exposure to microbial stimuli in early life programs the immune system towards Th2-type allergic response as described by 'hygiene hypothesis'.In allergic disorders there is shift of the Th1/Th2 cytokine balance towards a Th2 response, and causes the release of Interleukin-4, interleukin-5 and interleukin-13 as well as Immunoglobulin E production.

The diagnosis of AD is mainly clinical as there is no specific test for AD. Diagnosis of AD is based on specific a criterion which includes patient's history, clinical presentations as well as family history. In 1980 Hanifin and Rajka proposed major and minor diagnostic criteria based on clinical symptoms of AD. Williams coordinated a UK working party to attempt to simplify and refine the criteria given by Hanifin and Rajka in 1994. Severity of disease is evaluated by using widely accepted SCORing Atopic Dermatitis (SCORAD), based on extent of area involved, severity of symptoms and intensity of the subjective symptoms of pruritus and sleep disturbances.The chronic and recurrent nature of AD negatively impacts the quality of life (QOL) of patients as well as their family members. The symptoms of AD limit patient's physical, psychosocial development and quality of sleep.

The main goals of treatment are to improve the skin barrier function and hydration, to suppress inflammation and to control microbial colonization. It can be achieved through emollients, topical corticosteroids and topical calcineurin inhibitor like tacrolimus. Oral drugs like corticosteroids, methotrexate and cyclosporine are reserved for severe cases.

Probiotics are defined by World Health Orgnization as "live microorganisms, which when consumed in adequate amounts, confer a health effect on the host."Under the hypothesis that probiotics have global allergy protective effect, they have been extensively used for several conditions like inflammatory bowel disease, bronchial asthma and other allergic diseases. If children who are genetically predisposed to AD are supplemented with probiotics early in their life, series of events like antigenic competition, immune regulation and stimulation of innate immunity will occur, all of which might minimize their susceptibility to allergic disorders. Hence, investigators planned this study to see its role in AD.

Statement of problem and rationale:

The rationale for this therapeutic option is based on well-established effects of bacteria on cellular immune responses. The probiotics has an immunomodulatory property that plays an essential role in the development of normal immune tolerance. Early life exposure to these microbial agents plays an important role in maturation of Type 1 helper cell (Th1) immune responses and could inhibit development of allergic Type 2 helper cell (Th2) responses and IgE antibody production. Therefore the onset of AD could be prevented by probiotics and this treatment strategy could also be effective even when AD is already established.

In a meta-analysis conducted in 2017, involving 13 randomized controlled trials (RCT) with 1,070 children, significant difference in SCORAD values favoring probiotics over the control group was observed. Though, a high degree of heterogeneity was observed across these 13 trials.

Cochrane review, 2018 which included 39 RCTs found that probiotic treatment may slightly reduce SCORAD value. However the researcher concluded that the differences were not clinically significant. Recent review in 2019 on "prebiotics and probiotics in atopic dermatitis" based on various RCT and meta-analysis support the supplementation of probiotics for at least 8 weeks in improving severity score of AD.

Investigators have observed conflicting results of different studies with some showing significant advantages while some studies revealing no benefit. Almost all of the studies have suggested further research in different populations. Therefore, we are conducting this study to find out the effect of probiotics in AD in our institute.

OBJECTIVES

1. Primary objective: To investigate the efficacy of oral probiotics in the clinical outcome of Atopic dermatitis based on the SCORAD index
2. Secondary objectives: To find out the total duration of topical corticosteroid use in the interventional and conventional group.

To assess the impact of AD in children's family members based on FDLQI (Family Dermatology Life Quality Index)

MATERIALS AND METHODS Type of study design: Assessor blinded, randomized controlled trial. Setting: Hospital (Dermatology Outpatient Department, BPKIHS, Dharan). The probable duration of the study will be one year after approval from the Institutional Review Committee and Nepal Health Research Council (NHRC). Ethical Clearance: taken from the Institutional Review Committee (IRC), BPKIHS, and Nepal Health Research Council (NHRC).

Calculation of the sample size: According to a study done by Ekaputri et.al, it is reported that mean± SD of SCORAD index after intervention in probiotic group and control group was (18.09 ± 8.59) and (23.21± 8.71) respectively. Considering the least difference, 5.12 and pooled SD- 8.65, the sample size has been calculated at 95% CI and 80% power, using two means formula.

n = 44.56, adding 10% in calculated value for lost to follow-up, final sample size is 45 in each group. Thus a total of 98 patients will be enrolled.

n = 2σ2 (Z α/2 + Z β) 2 (μ1- μ2) 2

n= sample size of each group. σ = standard deviation 8.65 Z = reliability coefficient. 1.96 α = significance level. 0.05 Zβ= at 20% power 0.84 μ1 = mean (Probiotic) 18.09 μ2 = mean (Control) 23.21 d = mean difference 5.12

Randomization and allocation concealment:

A block randomization list will be generated with the block sizes 4, 6 and 8. Two parallel groups (1:1 ratio) of patients following computerized randomization will be produced. Prior to the enrollment of the patients a sequentially generated number with the treatment group will be written in sealed envelope, which will be prepared by independent dermatologist.

Interventional and conventional groups:

Interventional group: Children with AD meeting eligibility criteria receiving probiotics and conventional treatment (topical corticosteroid, topical tacrolimus, an oral antihistamine and emollients) Conventional group: Children with AD meeting eligibility criteria, under conventional treatment only.

Follow up:

Each patient will be asked for their follow up at 2, 4, 6, 8, 10 and 12 weeks of commencing treatment. In each follow up, every patient will be evaluated for the side effects and compliance to treatment. SCORAD index will be measured at baseline and at 4, 8, 10 and 12 weeks. FDLQI will be measured at baseline and at 8 weeks. Parents will be provided a card to record for flare of symptoms; total days of steroid use for the same and total flare episode will be recorded during 12 weeks follow up. Flare is defined as worsening of clinical features leading to use of corticosteroids for at least 3 consecutive days.

Family dermatology life quality index:

Parents or guardian of each children will be asked to fill the questionnaire intended to measure quality of life of family members whose relative have dermatological conditions. The standardized nepali version of FDLQI (MKA Basra, AY Finlay. Cardiff University 2005) will be used. Questions concern the influence of disease on parents QOL in the last month. Each question can be answered by selecting 1 out of 4 answers scored 0-3. The maximum score is 30 points and minimum 0 point. The higher the score lower the parents QOL.

Severity Index (SCORAD) It uses the rule of nine to assess extent of disease and evaluates five clinical characteristics to determine disease severity: i) erythema, ii) edema/ papulation, iii) oozing/crusts, iv) excoriation and v) lichenification. It also assesses subjective symptoms of pruritus and sleep loss with Visual Analogue Scales (VAS).

Based on SCORAD score, AD is categorized as

* Mild AD (SCORAD <25)
* Moderate (SCORAD 25-50)
* Severe (SCORAD >50)

Statistical Analysis:

Statistical analysis will be conducted both per protocol and intention to treat population (defined as all enrolled children to whom study drug will be given; with the last observation carried forward) basis using two sided tests.

Statistical methods proposed:

1. Descriptive statistics will be summarized as mean, median, percentage, standard deviation (SD) and interquartile range along with appropriate graphical and tabular presentation.
2. Intragroup SCORAD index and FDLQI score will be compared by paired t-test and between the groups by independent t- test.
3. In case of nonparametric data Mann- Whitney U test for independent groups and Wilcoxon signed- rank test for paired group will be used.
4. Chi-square test will be used to compare the categorical data. All statistical tests will be carried out at a significance level P<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Children with a diagnosis of atopic dermatitis that meet Hanifin and Rajka criteria
2. SCORAD ( SCORing Atopic Dermatitis) index 15- 50 at the time of enrollment

Exclusion Criteria:

1. SCORAD (SCORing Atopic Dermatitis) index <15 or >50.
2. Children treated with systemic corticosteroids, methotrexate, or cyclosporine in the previous 3 months and antibiotics in the previous 2 weeks.
3. Immunocompromised children.
4. Concomitant diagnosis of intolerance to gluten and/ or lactose.
5. Pre-existing hypersensitivity to components contained in the probiotics.
6. Children suffering from chronic infectious diseases.
7. A child with other known systemic diseases (heart, liver or kidney diseases).
8. Known case of short gut syndrome.
9. Refusal of children's parents to participate in the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants in each sex group | At the time of enrollment
  Sex distribution of Atopic Dermatitis patients in male, female or others group
Duration | At the time of enrollment
  Duration of Atopic Dermatitis
History Of Atopy | Enrollment
  Personal or Family history of atopy
Change in SCORing Atopic Dermatitis (SCORAD) index | Enrollment, 4 weeks, 8 weeks, 10 weeks and 12 weeks of treatment
  Based on three aspects, extent of disease, disease severity and subjective symptoms combine to give a maximum possible score of 103.

SECONDARY OUTCOMES:
Number of participants having each of systemic illnesses | Enrollment
  Systemic diseases like heart, liver and kidney diseases
Number of participants who had taken past treatment | Enrollment
  Different types of treatment received -either medicinal or traditional
Age of Onset | Enrollment
  Age of onset of Atopic Dermatitis
Change in Family Dermatology Life Quality Index | At the time of enrollment and at 8 weeks of commencing treatment.
  It will be measured using a standard Nepali version of Family Dermatology Life Quality Index questionnaire. Questions concern the influence of disease on parents QOL in the last month. Each question can be answered by selecting 1 out of 4 answers scored 0-3. The maximum score is 30 points and minimum 0 point. The higher the score lower the parents Quality of Life.

CONTACTS AND LOCATIONS:
Locations (1):
- B.P. Koirala Institute of Health Sciences, Dharān, Nepal

IPD SHARING:
Plan to Share IPD: No